CLINICAL TRIAL: NCT00950703
Title: Primary Care Audit of Global Risk Management
Acronym: PARADIGM
Status: Completed | Type: Observational
Sponsor: Canadian Collaborative Research Network (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Milan Gupta, MD, Canadian Collaborative Research Network
Other Study IDs: D3560L00086
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Diseases
Keywords: Assessing the perceptions of Canadian Primary care physicians towards global Cardiovascular risk assessment.
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Assessing the perception of Canadian Primary Care Physicians towards global cardiovascular risk assessment.
2. Correlating physician perceptions to actual practice data, gathered via a retrospective chart audit.
3. Evaluating the impact of a prospective educational and peer-practice pattern intervention on future assessment o cardiovascular risk and
4. Assessing the role of carotid atherosclerosis assessment(Carotid IMT and plaque) as an adjunct to global risk prediction.

DETAILED DESCRIPTION:
The majority of cardiovascular events occur in people with low to intermediate Framingham Risk Score. Despite evidence-based guidelines, the appropriate use of lipid-lowering therapies in this population remains limited and controversial. Strategies to refine risk stratification in primary prevention have been poorly adopted. Dissemination of practice-changing trials and closing the care gap in primary care remain a priority and a challenge. Considerable confusion remains regarding the optimal application of lipid-lowering therapy in primary prevention. Importantly, it remains largely unknown which tools or techniques are used by Canadian primary care physicians to identify global vascular risk, and what barriers exist to implementing risk reduction therapies in such individuals.

For primary prevention of patients with normal levels of LDL-Cholesterol who are at increased risk on the basis of elevated hsCRP, it remains unproven whether statin therapy will effectively reduce vascular event rates. The JUPITER trial was launched in 2003 comparing rosuvastatin with placebo in 18,000 primary prevention patients with LDL-cholesterol of less than 3.36mM who also have an hsCRP of greater than 2 mg/L. This trial has been stopped early due to unequivocal morbidity and mortality benefits in favor of the treatment strategy, and the final results will be available in early November, 2008. JUPITER, once published, will require a major change in physician behavior with respect to screening and treating cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

1. Men more than or equal to 40 yrs old and women more than or equal to 50 yrs old;
2. No previous history of atherosclerosis( angina, TIA, myocardial infarction, stroke, peripheral arterial disease);
3. Non-diabetic;
4. Absence of lipid lowering treatment (current or past).

Exclusion Criteria:

1. Known history of atherosclerosis or diabetes;
2. Use of lipid lowering therapies (statins, ezetimibe, fibrates, niacin, fish oil);
3. Use of postmenopausal hormone replacement therapy;
4. Use of immunosuppressant's or steroids;
5. Active liver disease or hepatic dysfunction(ALT>2times the ULN);
6. Active renal disease (baseline Creatinine >170 umol/L);
7. History of malignancy within the past 5-years;
8. Chronic inflammatory conditions such as arthritis, lupus or inflammatory bowel disease;
9. Known alcohol or drug abuse;
10. Failure to provide informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinics.
Sampling Method: Probability Sample
Enrollment: 3015 (Actual)
Dates: Start 2009-03; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The Primary objective of the PARADIGM study is to evaluate the impact of an educational and peer-practice pattern intervention on primary care physician behavior towards global cardiovascular risk prediction in otherwise healthy individuals. | 1 year

SECONDARY OUTCOMES:
Evaluate the prevalence of classic and novel markers of risk (hsCRP and ApoB/ApoA1). | 1 year
Evaluate within a sub-study, the feasibility of carotid atherosclerosis assessment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Milan K Gupta, MD, Principal Investigator — Canadian Collaborative Research Network; Subodh Verma, MD, Principal Investigator — Canadian Collaborative Research Network
Locations (1):
- CCRN, Brampton, Ontario, Canada

REFERENCES:
- [Derived] Law TK, Yan AT, Gupta A, Kajil M, Tsigoulis M, Singh N, Verma S, Gupta M. Primary prevention of cardiovascular disease: global cardiovascular risk assessment and management in clinical practice. Eur Heart J Qual Care Clin Outcomes. 2015 Jul 1;1(1):31-36. doi: 10.1093/ehjqcco/qcv002. PMID 29474565